CLINICAL TRIAL: NCT06641570
Title: Effects of a Land and Aquatic Exercise-based Program on Pain, Mobility and Quality of Life in Patients With Chronic Low Back Pain: A Randomized Controlled Trial
Brief Title: Effects of a Land and Aquatic Exercise-based Program on Pain, Mobility and Quality of Life in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Leiria (Other)
Collaborators: Instituto PolitÃ©cnico de Castelo Branco (Unknown)
Responsible Party: Principal Investigator, Joana Catarina Carvalho Borges, Principal Investigator, Instituto Politécnico de Leiria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE/IPLEIRIA/47/2024
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-01

CONDITIONS: Chronic Low-back Pain (cLBP)
Keywords: Pain; Exercise; Hydrotherapy; Aquatic Therapy; Disability
MeSH Terms: conditions — Pain; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aquatic Exercise Program + Land-exercise Program (Experimental): This intervention will include 8 sessions in 8 weeks, once a week. Each session will last between 25 to 35 minutes and will be divided into two components: core stability exercises and stretching of the trunk and lower limbs.
  Core Stability Exercises: These will consist of isometric exercises maintained for 7-8 seconds, 8-12 repetitions, 1 set, with brief rest intervals of 3 seconds between repetitions and 30 seconds to 1 minute between exercises. Exercises will include abdominal hollowing, side bridge (both sides), supine extension bridge, lower limb extension from prone (both sides), and alternate arm and leg raise from quadruped.
  Stretching Exercises: Participants will perform muscle stretching exercises, holding the maximum stretch for 30 seconds to 1 minute, and returning to the original position, followed by 5 to 10 seconds of rest. Each exercise will be repeated two to three times. Stretches will target the hamstrings, iliopsoas, piriformis, and tensor fasciae latae.
  Interventions: Other: Aquatic Exercise Program; Other: Land-based Exercise Program
- Aquatic Exercise Program (Active Comparator): This intervention will include 16 sessions of an aquatic-exercise program, twice a week, over 8 weeks at a water temperature between 32-34°C. Each session will be conducted in groups of 8 to 12 patients and will last about 45 minutes.
  The aquatic exercise sessions will include a warm-up phase: walking forwards, sideways, and backwards; a training phase: active range of motion exercises for the spine, upper and lower limbs; aerobic exercises with jumps and static running at various speeds; muscle strengthening, 8-12 repetitions, 1-2 sets, 8-10 exercises including hip flexion, extension, adduction, and abduction, knee flexion and extension, knee cycling, shoulder flexion, extension, and abduction, elbow flexion, extension, and pronation-supination, squatting, and stretching exercises for the neck, trunk, and limbs; and a relaxation/cool-down phase: including lying supine and low-impact exercises such as slow walking, squatting, and standing.
  Interventions: Other: Aquatic Exercise Program

INTERVENTIONS:
Other: Aquatic Exercise Program — This intervention will include 16 sessions of an aquatic-exercise program, twice a week, over 8 weeks at a water temperature between 32-34°C. Each session will be conducted in groups of 8 to 12 patients and will last about 45 minutes.
Other: Land-based Exercise Program — This intervention will include 8 sessions in 8 weeks, once a week. Each session will last between 25 to 35 minutes and will be divided into two components: core stability exercises and stretching of the trunk and lower limbs.
  Arms: Aquatic Exercise Program + Land-exercise Program

SUMMARY:
The goal of this randomized clinical trial] is to study the effect of a combined aquatic and land-based exercise program compared to an aquatic program on pain, functional disability, and quality of life in adults with chronic low back pain. The main question it aims to answer is: "Does a combined aquatic and land-based exercise program improve functional disability and quality of life and reduce pain in adults with chronic low back pain?".

Participants will perform an aquatic exercise program (control group) or a combined aquatic and land-based exercise program (experimental group).

Researchers will compare groups to find any differences in pain, funcional disability and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Both gender;
* Portuguese nationality;
* Aged over 18 years;
* Chronic Low Back Pain lasting three months or longer and with an intensity of 3 or higher on the Visual Analogue Scale at rest.

Exclusion Criteria:

* Individuals who refuse to participate or do not provide informed consent;
* Pain radiating to the lower limb;
* Recent pregnancy or childbirth (less than 8 weeks ago);
* Ongoing physical therapy treatments;
* Severe rheumatological, neurological, neoplastic, cardiovascular diseases or other conditions that could prevent full participation in the intervention;
* History of spinal surgery;
* Inflammatory, infectious, or malignant spinal diseases;
* Psychiatric disorders that may affect adherence and symptom assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Pain | From enrollment to the end of treatment at 8 weeks
  Quantitive variable evaluated with Visual Analogue Scale (Minimum: 0; Maximum 10). Higher values correspond to worse outcome.
Functional Disability | From enrollment to the end of treatment at 8 weeks
  Quantitive variable evaluated with Oswestry Disability Index - version 2.0. (Minimum: 0; Maximum 100). Higher values correspond to worse outcome.
Quality of life | From enrollment to the end of treatment at 8 weeks
  Quantitive variable evaluated with MOS Short Form Health Survey 36 Item v2. (Minimum: 0; Maximum 100). Higher values correspond to better outcome.

SECONDARY OUTCOMES:
Lumbar spine range of motion | From enrollment to the end of treatment at 8 weeks
  Quantitive variable evaluated with Modified-Modified Schober Test.
Fear of movement or (re)injury | From enrollment to the end of treatment at 8 weeks
  Quantitive variable evaluated with Tampa Scale of Kinesiophobia-13. (Minimum: 13; Maximum 52). Higher values correspond to worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Joana Borges, PT, Principal Investigator — Instituto Politécnico de Leiria; Diogo Monteiro, PhD, Study Director — Instituto Politécnico de Leiria; Pedro Mendes, PhD, Study Director — Instituto Politécnico de Castelo Branco
Locations (1):
- Polytechnic Institute of Leiria, Leiria, Leiria District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borges J, Monteiro D, Silva FM, Jacinto M, Pastilha T, Duarte-Mendes P. Effects of a land and aquatic exercise-based program on pain, mobility and quality of life in patients with chronic low back pain: a study protocol for a randomized controlled trial. PLoS One. 2025 May 20;20(5):e0320858. doi: 10.1371/journal.pone.0320858. eCollection 2025. PMID 40392887